CLINICAL TRIAL: NCT01077401
Title: Ranibizumab for Edema of the Macula in Diabetes: Protocol 3 With High Dose - the READ 3 Study
Acronym: READ 3
Status: Completed | Phase: Phase 2 | Type: Interventional
Sponsor: Johns Hopkins University (Other)
Collaborators: Juvenile Diabetes Research Foundation (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Treatment
Other Study IDs: NA_00034586
Record Dates: First submitted 2010-02-26; First posted 2010-03-01 (Estimated); Results first posted 2017-04-28 (Actual); Last update posted 2017-04-28 (Actual); Status verified 2017-03

CONDITIONS: Diabetic Macular Edema
Keywords: Diabetic; edema; DME
MeSH Terms: conditions — Edema | interventions — Ranibizumab

STUDY DESIGN:
Who Masked: Participant
Oversight: Data Monitoring Committee: Yes

ARMS (2):
- Ranibizumab 0.5mg (Experimental): Intravitreal injections of ranibizumab 0.5mg dose for six monthly treatments then additional treatments with ranibizumab 0.5mg dose if the subject meets re-treatment criteria.
  Interventions: Drug: Ranibizumab
- Ranibizumab 2.0 mg (Experimental): Intravitreal injections of ranibizumab 2.0 mg dose for six monthly treatments then additional treatments with ranibizumab 2.0 mg dose if the subject meets re-treatment criteria.
  Interventions: Drug: ranibizumab

INTERVENTIONS:
Drug: Ranibizumab — Intravitreal injections of ranibizumab 0.5mg dose for six monthly treatments then additional treatments with ranibizumab 0.5mg dose if the subject meets re-treatment criteria.
  Other Names: lucentis
  Arms: Ranibizumab 0.5mg
Drug: ranibizumab — Intravitreal injections of ranibizumab 2.0 mg dose for six monthly treatments then additional treatments with ranibizumab 2.0 mg dose if the subject meets re-treatment criteria.
  Other Names: lucentis high-dose
  Arms: Ranibizumab 2.0 mg

SUMMARY:
The purpose of this study is to investigate the safety, tolerability, bioactivity, and dose response of two different dosages (0.5 mg and 2.0 mg) of ranibizumab (RBZ) in patients with diabetic macular edema (DME).

ELIGIBILITY:
Inclusion Criteria:

Signed informed consent and authorization of use and disclosure of protected health information

* Age ≥18 years
* Diagnosis of diabetes mellitus (type 1 or type 2)
* Serum HbA1c ≥ 5.5% within 12 months of randomization. Retinal thickening secondary to diabetes mellitus (diabetic macular edema) involving the center of the fovea
* Diagnosis must be confirmed by fluorescein angiography and OCT images
* Foveal thickness of ≥ 250 μm,
* Best corrected visual acuity score in the study eye of 20/40 to 20/320 inclusive (Snellen equivalents using the ETDRS protocol at a distance of 4 meters). The non-study eye must be ≥ 20 letters (approximate Snellen equivalent 20/400).
* In the opinion of the investigator, decreased vision in the study eye is due to foveal thickening from DME and not from other obvious causes of decreased vision If a female of childbearing potential, a negative pregnancy test and commitment to the use of at least two forms of effective contraception (birth control) for the duration of the study are necessary.

Exclusion Criteria:

* Panretinal photocoagulation or macular photocoagulation within 3 months of study entry in the study eye
* Use of intraocular or periocular injection of steroids in the study eye (e.g., triamcinolone) within 3 months of study entry
* Previous participation in a study and receipt of anti-angiogenic drugs (pegaptanib sodium, ranibizumab, bevacizumab, anecortave acetate, protein kinase C inhibitor, etc.) within 2 months of study entry
* Proliferative diabetic retinopathy in the study eye, with the exceptions of
* Inactive, fibrotic proliferative diabetic retinopathy that has regressed following panretinal laser photocoagulation OR
* Tufts of neovascularization elsewhere (NVE) less than one disc area with no vitreous hemorrhage
* Vitreomacular traction or epiretinal membrane in the study eye evident biomicroscopically or by optical coherence tomography (OCT)
* Structural damage to the center of the macula in the study eye likely to preclude improvement in visual acuity following the resolution of macular edema, including atrophy of the retinal pigment epithelium, subretinal fibrosis, laser scar(s), macular ischemia, or organized hard exudate plaque
* Ocular disorders in the study eye that may confound interpretation of study results, including retinal vascular occlusion, retinal detachment, macular hole, or choroidal neovascularization of any cause (e.g., age related macular degeneration (AMD), ocular histoplasmosis, or pathologic myopia)
* Concurrent disease in the study eye that could compromise visual acuity or require medical or surgical intervention during the first 6-month study period
* Cataract surgery in the study eye within 3 months of study entry; Yttrium-Aluminum- Garnet (YAG) laser capsulotomy within 1 month of study entry; or any other intraocular surgery within 3 months preceding Day 0.
* History of vitreoretinal surgery in the study eye within 3 months of study entry
* Uncontrolled glaucoma (defined as intraocular pressure ≥30 mm Hg despite treatment with anti-glaucoma medications)
* Blood pressure exceeding 180/100 (sitting) during the screening period
* Uncontrolled diabetes mellitus, as evidenced by glycosylated hemoglobin (HbA1c) value >13%
* Renal failure requiring dialysis or renal transplant
* Premenopausal women unwilling to commit to adequate contraception
* History of other diseases, metabolic dysfunction, physical examination finding, or clinical laboratory finding giving reasonable suspicion of a disease or condition that contraindicates the use an investigational drug, might affect interpretation of the results of the study, or render the subject at high risk from treatment complications
* International normalized ratio (INR) ≥ 3.0 (e.g. due to current treatment with warfarin). The use of aspirin or other anticoagulants is not an exclusion
* History of cerebral vascular accident, myocardial infarction, transient ischemic attacks within 3 months of study enrollment.
* Have a history of hypersensitivity to ranibizumab or any of its components
* Have the presence of active malignancy, including lymphoproliferative disorders. Subjects with a history of fully resolved basal or squamous cell skin cancer may be enrolled.

Other

* Inability to comply with study or follow-up procedures
* Any other condition that the investigator believes would pose a significant hazard to the subject if the investigational therapy were initiated.
* Participation in another simultaneous medical investigation or trial

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 152 (Actual)
Dates: Start 2010-02; Primary Completion 2012-03 (Actual); Study Completion 2013-03 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Diana V Do, MD, Principal Investigator — Truhlsen Eye Institute, University of Nebraska Medical Center
Locations (13):
- United States (13):
  - Retina Vitreous Associates, Beverly Hills, California
  - University of California San Diego, La Jolla, California
  - Doheny Eye Institute, Los Angeles, California
  - East Bay Retina Institute, Oakland, California
  - Retina Macula Institute, Torrance, California
  - Retina Group of Florida, Fort Lauderdale, Florida
  - Retina Institute of Hawaii, Honolulu, Hawaii
  - Illinois Retina Associates, Joliet, Illinois
  - University of Kansas, Prairie Village, Kansas
  - Johns Hopkins University Wilmer Eye Institute, Baltimore, Maryland
  - Eye Care Specialists, Kingston, Pennsylvania
  - Black Hills Eye Institute, Rapid City, South Dakota
  - Texas Retina Associates, Arlington, Texas

RESULTS

PARTICIPANT FLOW:
Period: Overall Study
Arm/Group | Ranibizumab 0.5mg | Ranibizumab 2.0 mg
Started | 77 | 75
Completed | 59 | 54
Not Completed | 18 | 21

BASELINE CHARACTERISTICS:
Groups:
- Total: Total of all reporting groups
Arm/Group | Ranibizumab 0.5mg | Ranibizumab 2.0 mg | Total
Number analyzed (Participants) | 77 | 75 | 152
Age, Continuous [Mean (Full Range); unit: years] | 64.8 [35 to 87] | 63.5 [48 to 84] | 64.1 [35 to 87]
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 30 | 37 | 67
  Male | 47 | 38 | 85
Race (NIH/OMB) [Count of Participants; unit: Participants]
  American Indian or Alaska Native | 0 | 0 | 0
  Asian | 4 | 5 | 9
  Native Hawaiian or Other Pacific Islander | 0 | 0 | 0
  Black or African American | 6 | 13 | 19
  White | 45 | 39 | 84
  More than one race | 0 | 0 | 0
  Unknown or Not Reported | 22 | 18 | 40
Region of Enrollment [Number; unit: participants]
  United States | 77 | 75 | 152

OUTCOME MEASURES:

1. Primary Outcome: Deaths Due to Myocardial Infarction
Time Frame: 6 Months
Measure: Number; unit: participants
Arm/Group | Ranibizumab 0.5mg | Ranibizumab 2.0 mg
Number analyzed (Participants) | 77 | 75
participants | 1 | 3

2. Secondary Outcome: Mean Change in Best Corrected Visual Acuity From Baseline to Month 6
Description: Mean change in best corrected visual acuity (BCVA) (ETDRS) at 4 meters in the study eye over time through month 6.
Time Frame: baseline 6 Months
Measure: Mean (Standard Deviation); unit: letters
Arm/Group | Ranibizumab 0.5mg | Ranibizumab 2.0 mg
Number analyzed (Participants) | 77 | 75
letters | 9.34 (10.34) | 7.04 (8.33)

3. Secondary Outcome: Mean Change in Retinal Thickness at Month 6
Time Frame: baseline to6 Months
Population: Data was not collected for 4 participants in the Ranibizumab 0.5mg group for this outcome measure.
Measure: Mean (Standard Deviation); unit: µm
Arm/Group | Ranibizumab 0.5mg | Ranibizumab 2.0 mg
Number analyzed (Participants) | 73 | 75
µm | 168.57 (145.67) | 159.69 (124.50)

ADVERSE EVENTS:
Time Frame: 6 months
Arm/Group | Ranibizumab 0.5mg | Ranibizumab 2.0 mg
Serious Adverse Events (participants affected / at risk) | 1/77 | 3/75
Other Adverse Events (participants affected / at risk) | 1/77 | 0/75
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Ranibizumab 0.5mg (N=77) | Ranibizumab 2.0 mg (N=75)
Deaths from Myocardial Infarction within 6 months of starting study (Cardiac disorders) | 1 (1) | 3 (3)
OTHER ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Ranibizumab 0.5mg (N=77) | Ranibizumab 2.0 mg (N=75)
Loss of 30 or more letters (Eye disorders) | 1 (1) | 0 (0)

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: No